CLINICAL TRIAL: NCT00233623
Title: A Randomised, Non-Comparative, Multicentre, Phase II, Parallel-Group Trial Of ZD1839 (Iressa™) In Combination With 5 Fluorouracil, Leucovorin And Cpt-11 (Irinotecan) In Patients With Metastatic Colorectal Cancer
Brief Title: Irinotecan, 5-Fluorouracil and Leucovorin With or Without Iressa in the Treatment of Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0138
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Gefitinib; Irinotecan; Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: Iressa (Gefitinib)
Drug: Irinotecan
Drug: 5Fluorouracil
Drug: Leucovorin

SUMMARY:
The aim of the study is to determine if Iressa added to chemotherapy with Irinotecan, 5Fluorouracil and Leucovorin can prolong the period of time without any disease worsening (Time to Progression) in patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic colorectal cancer
* Presence of measurable metastases
* No previous treatment for metastatic cancer

Exclusion Criteria:

* No presence of Central Nervous System metastases
* No other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190
Dates: Start 2004-07; Primary Completion 2006-01 (Estimated); Study Completion 2006-01 (Estimated)

PRIMARY OUTCOMES:
Time to progression (6 months after Last patient in)

SECONDARY OUTCOMES:
Objective Response Rate, Duration of Response, Disease control rate, Overall Survival, (6 months after Last patient in)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Italy Medical Director, MD, Study Director — AstraZeneca
Locations (13):
- Italy (13):
  - Research Center, Bari
  - Research Site, Bergamo
  - Research Site, Catania
  - Research Site, Cremona
  - Research Site, Cuneo
  - Research Site, La Spezia
  - Research Site, L’Aquila
  - Research Site, Milan
  - Research Site, Palermo
  - Research Site, Pescara
  - Research Site, Rozzano
  - Research Site, Torino
  - Research Site, Venezia